CLINICAL TRIAL: NCT03737630
Title: Effects of Inspiratory Muscle Training in Individuals Who Have Cystic Fibrosis
Brief Title: Inspiratory Muscle Training in Individuals With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Patri-cia Angelica de Miranda Silva Nogueira, PhD, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1a2b3c4d5e
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; quality of life; posture
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GExp (Experimental): This group will perform the inspiratory muscle training with moderate load
  Interventions: Device: Inspiratory muscle training
- GCon (Active Comparator): This group will initiate inspiratory muscle training with low load
  Interventions: Device: Inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — This group will initiate inspiratory muscle training with 40% of the MIP load and each week will have a load increase of 10% of the initial MIP up to 4 weeks of training

SUMMARY:
Cystic fibrosis is a genetic disease that affects some organs of the human body. Among them, the lungs tend to be the most affected due to the accumulation of mucus in the airways, which in addition to avoiding the passage of air, favors pulmonary infections. With the evolution of the condition, secondary complications arise, such as postural changes, decreased respiratory muscle strength, decreased functional capacity and, consequently, quality of life. Therefore, respiratory muscle training may be an intervention that improves the respiratory condition of these individuals, allowing an improvement in the quality of life and may delay the evolution of respiratory symptoms. Thus, this study aims to investigate a home protocol of respiratory muscle training on respiratory muscle strength, lung function, quality of life, posture and functional capacity in adolescents and adults with cystic fibrosis. The researchers believe that the training can cause an improvement in the studied variables, and can be inserted in the usual treatment of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis, confirmed by the sweat test;
* 14 - 25 years;
* Clinical stability;
* Absence of bacterial colonization for 4 weeks;
* Both sexes;

Exclusion Criteria:

* Inability to perform the protocol established by the study;
* Present any intercurrence during data collection;
* Being unable to understand and / or perform procedures.
* Colonization during study participation;
* Patient hospitalization due to worsening of the clinical picture.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Posture at 4 weeks | Baseline and after 4 weeks of training
  Inclinometer Danoplus®
Change from baseline Health-related quality of life at 4 weeks | Baseline and after 4 weeks of training
  Health-related quality of life questionnaire (HRQoL)

SECONDARY OUTCOMES:
Change from baseline Respiratory muscle strength at 4 weeks | Baseline and after 4 weeks of training
  MVD300®
Change from baseline Pulmonary function at 4 weeks | Baseline and after 4 weeks of training
  Spirometry test using Koko® device
Change from baseline Functional capacity at 4 weeks | Baseline and after 4 weeks of training
  three-minute step test

CONTACTS AND LOCATIONS:
Overall Officials: Victor Oliveira, Master, Study Chair — Universidade Federal do Rio Grande do Norte
Locations (1):
- Universidade Federal do Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stanford G, Ryan H, Solis-Moya A. Respiratory muscle training for cystic fibrosis. Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD006112. doi: 10.1002/14651858.CD006112.pub5. PMID 33331663